CLINICAL TRIAL: NCT01049074
Title: A Random Controlled Test (RCT): Acupuncture Treatment on Nonspecific Low Back Pain (NLBP) (ANLBP)
Brief Title: A Random Controlled Test (RCT): Acupuncture Treatment on Nonspecific Low Back Pain (NLBP)
Acronym: ANLBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Wang LinPeng / Director of Acupuncture Department, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JKH 081
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2008-11

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Acupuncture; RCT
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verus acupuncture (Experimental)
  Interventions: Other: Acupuncture Treatment
- Sham acupuncture (Sham Comparator)
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture Treatment — Acupuncture is a technique of inserting and manipulating fine needles into specific points on the body to relieve pain or for therapeutic purposes.
  Arms: Verus acupuncture
Other: Sham acupuncture — Sham acupuncture is inserting needles superficially, without manipulating, into specific points on the body.
  Arms: Sham acupuncture

SUMMARY:
Hypothesis: Acupuncture procedure of He's Santong Methods could be an option to treat nonspecific low back pain.

DETAILED DESCRIPTION:
He's Santong Methods is a combined manipulated needling methods, including filiform needling, fire needling and bloodletting needling, which was created by Dr. He Puren who is one of the most famous TCM doctors in China.

ELIGIBILITY:
Inclusion Criteria:

* The patient who is suffering the Non-specific Low Back Pain which meets the diagnostic criterion of posterior ramus of lumbar spinal nerve syndrome.
* The patient who is from 18 to 79 years old.
* The patient who can comprehensively understand and fill in the questionnaires about the disease.
* The patient who suffered problems no less than 12 weeks.
* The patient who have not the other diseases which can result in back pain.
* The patient who received the clear examinations of X-ray, CT scan or MRI.
* The patient who wrote the informed consents.

Exclusion Criteria:

* The patient whose low back pain is the consequences of spondyloschisis, Spondylolysis, osteoarthritis, osteoporosis, internal disease, metastatic tumor.
* The patient who have the hemorrhagic disease such as hemophilia.
* The patient who have the spinal diseases which have not been diagnosed clearly.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Score of SF-36 | 4 weeks, 8 weeks, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 4 weeks, 8 weeks, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linpeng Wang, M.D., Study Chair — Beijing TCM Hospital; Stratulat Ioan Sorin, M.D., Principal Investigator — Hospital CF Iasi, Clinic of Rehabilitation Medicine, Phys. Med., Balneoclimatology
Locations (2):
- Beijing TCM Hospital, Beijing, Beijing Municipality, China
- Hospital CF Iasi, Clinic of Rehabilitation Medicine, Phys. Med., Balneoclimatology, Lasi, Romania